CLINICAL TRIAL: NCT02460614
Title: Comparison Between Rhinopharyngeal Retrograde Clearance and Nasopharyngeal Aspiration in Children With Acute Viral Bronchiolitis
Brief Title: Effects of Rhinopharyngeal Retrograde Clearance in Children With Acute Viral Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marcio Vinicius Fagundes Donadio, Professor, Pontificia Universidade Católica do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRR-15
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Acute Viral Bronchiolitis
Keywords: bronchiolitis; respiratory physiotherapy; pediatrics; rhinopharyngeal clearance
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rhinopharyngeal clearance + 0.9% saline (Experimental): The retrograde rhinopharyngeal clearance (RRC) is based on the inspiratory reflex that follows a slow and prolonged expiration (passive exhalation technique performed using a slow thoracic-abdominal compression that begins at the end of a spontaneous exhalation and continues until the expiratory reserve volume). At the end of the expiratory time, the child's mouth was closed by the hand of the researcher (raising the lower jaw), leading the child to perform a nasal aspiration maneuver. The instillation of saline (0.9%) preceded this step, resulting in the inhalation of the substance during the forced inspiration, contributing to the nasopharyngeal clearance.
  Interventions: Procedure: Rhinopharyngeal clearance; Other: 0.9% saline
- Aspiration + 0.9% saline (Active Comparator): Nasopharyngeal aspiration consisted in the introduction of a catheter that, by using negative pressure (vacuum), promotes the suction of secretion from the airways. In order to do that, a sterile aspiration catheter was connected to an extension and carefully introduced into the nasal cavity of the patient. The saline instillation of 0.9% was used for humidification before the procedure.
  Interventions: Procedure: Aspiration; Other: 0.9% saline

INTERVENTIONS:
Procedure: Rhinopharyngeal clearance — At the end of the expiratory time, the child's mouth was closed by the hand of the researcher (raising the lower jaw), leading the child to perform a nasal aspiration maneuver.
  Arms: Rhinopharyngeal clearance + 0.9% saline
Procedure: Aspiration — A sterile aspiration catheter was connected to an extension and carefully introduced into the nasal cavity of the patient.
  Arms: Aspiration + 0.9% saline
Other: 0.9% saline — 0.9% saline consists of physiological solution and was instilled in both experimental groups.

SUMMARY:
The purpose of this study is to compare the immediate effects of retrograde rhinopharyngeal clearance with nasopharyngeal aspiration in children admitted with acute viral bronchiolitis. The investigators selected children, up to 12 months old, admitted for acute viral bronchiolitis. Patients were divided in aspiration group (AG), submitted to nasopharyngeal aspiration, and clearance group (CG), submitted to retrograde rhinopharyngeal clearance with physiological solution (0.9%) instillation (RRC) technique. In both groups children were evaluated three times in the same day in order to verify cardiorespiratory parameters, clinical score of respiratory dysfunction and adverse effects.

DETAILED DESCRIPTION:
Children up to 12 months old, admitted for acute viral acute viral bronchiolitis were selected. All children participating in the study should be in the first 48 hours of hospitalization. Patients were divided in aspiration group (AG), submitted to nasopharyngeal aspiration, and clearance group (CG), submitted to retrograde rhinopharyngeal clearance (RRC) technique with physiological solution (0.9%) instillation. In both groups children were evaluated three times in the same day (data collection 1 (C1) - performed early in the morning; data collecting 2 (C2) - performed in the early afternoon; and data collecting 3 (C3) - performed in the evening). In each data collection, cardiorespiratory parameters and clinical score of respiratory dysfunction were evaluated before procedures (T0), 10 minutes after (T1) and 30 minutes after (T2). Adverse effects were evaluated during the whole day of the study.

ELIGIBILITY:
Inclusion Criteria:

* acute viral bronchiolitis diagnosis
* indication for hospital admission

Exclusion Criteria:

* history of lung disease related to prematurity (bronchopulmonary dysplasia)
* heart diseases
* chronic lung diseases (cystic fibrosis)
* pneumonia
* unstable hemodynamic process (ARDS or sepsis)
* subcutaneous edema
* admission to the intensive care unit
* need for mechanical ventilation or tracheostomy
* neurological diseases

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of chest retractions as a measure of respiratory distress | 30 minutes
Occurrence of wheezing as a measure of respiratory distress | 30 minutes
Number of nasal bleeding events as a measure of adverse effects | 1 day
Number of vomit episodes as a measure of adverse effects | 1 day

SECONDARY OUTCOMES:
Measurement of the heart rate using an oximeter | 30 minutes
Measurement of the respiratory rate | 30 minutes
Measurement of the oxygen saturation using an oximeter | 30 minutes
Severity scores on the Wood clinical score | 30 minutes

REFERENCES:
- [Background] Gomes EL, Postiaux G, Medeiros DR, Monteiro KK, Sampaio LM, Costa D. Chest physical therapy is effective in reducing the clinical score in bronchiolitis: randomized controlled trial. Rev Bras Fisioter. 2012 Jun;16(3):241-7. doi: 10.1590/s1413-35552012005000018. Epub 2012 Apr 12. PMID 22499404
- [Background] Rochat I, Leis P, Bouchardy M, Oberli C, Sourial H, Friedli-Burri M, Perneger T, Barazzone Argiroffo C. Chest physiotherapy using passive expiratory techniques does not reduce bronchiolitis severity: a randomised controlled trial. Eur J Pediatr. 2012 Mar;171(3):457-62. doi: 10.1007/s00431-011-1562-y. Epub 2011 Sep 17. PMID 21927808
- [Background] Sanchez Bayle M, Martin Martin R, Cano Fernandez J, Martinez Sanchez G, Gomez Martin J, Yep Chullen G, Garcia Garcia MC. [Chest physiotherapy and bronchiolitis in the hospitalised infant. Double-blind clinical trial]. An Pediatr (Barc). 2012 Jul;77(1):5-11. doi: 10.1016/j.anpedi.2011.11.026. Epub 2012 Jan 26. Spanish. PMID 22281403
- [Background] Jacinto CP, Gastaldi AC, Aguiar DY, Maida KD, Souza HC. Physical therapy for airway clearance improves cardiac autonomic modulation in children with acute bronchiolitis. Braz J Phys Ther. 2013 Nov-Dec;17(6):533-40. doi: 10.1590/S1413-35552012005000120. Epub 2013 Nov 1. PMID 24271093
- [Background] Jarvis K, Pirvu D, Barbee K, Berg N, Meyer M, Gaulke L, Pate BM, Roberts C. Change to a standardized airway clearance protocol for children with bronchiolitis leads to improved care. J Pediatr Nurs. 2014 May-Jun;29(3):252-7. doi: 10.1016/j.pedn.2013.11.007. Epub 2013 Nov 27. PMID 24333327
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196
- [Derived] Gomes GR, Calvete FP, Rosito GF, Donadio MV. Rhinopharyngeal Retrograde Clearance Induces Less Respiratory Effort and Fewer Adverse Effects in Comparison With Nasopharyngeal Aspiration in Infants With Acute Viral Bronchiolitis. Respir Care. 2016 Dec;61(12):1613-1619. doi: 10.4187/respcare.04685. Epub 2016 Aug 23. PMID 27555618